CLINICAL TRIAL: NCT06468007
Title: SAP Version 28 May 2024. Comparative Effects of Methylprednisolone and Prednisolone on the Risk of Acute Decompensated Heart Failure - An Emulated Target Trial
Brief Title: Comparative Effects of Methylprednisolone and Prednisolone on the Risk of Acute Decompensated Heart Failure - An Emulated Target Trial
Status: Completed | Type: Observational
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SAP version 28 May 2024.
Record Dates: First submitted 2024-05-29; First posted 2024-06-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; With Decompensation
Keywords: Methylprednisolone; Prednisolone; Emulated target trial
MeSH Terms: conditions — Heart Failure | interventions — Methylprednisolone; Prednisolone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Methylprednisolone treatment group: Patients receiving 4 mg or 16 mg methylprednisolone tablets for any of the following conditions: Pulmonary, Rheumatology and musculoskeletal; Neurology and ophthalmology; Dermatology; Endocrinology and metabolic; Gastrointestinal; Hematology and immunology; Nephrology.
  Interventions: Drug: Methylprednisolone Tablet
- Prednisolone treatment group: Patients receiving 5 mg or 20 mg prednisolone tablets for any of the following conditions: Pulmonary, Rheumatology and musculoskeletal; Neurology and ophthalmology; Dermatology; Endocrinology and metabolic; Gastrointestinal; Hematology and immunology; Nephrology.

INTERVENTIONS:
Drug: Methylprednisolone Tablet — Patients receiving equipotent doses of methylprednisolone or prednisolone . Dosages will be determined at the discretion of the treating physician, customized for the specific clinical need in accordance with local guidelines.
  Other Names: Prednisolone Tablet
  Groups: Methylprednisolone treatment group

SUMMARY:
The investigators aim to emulate a target trial to compare the risk of acute decompensated heart failure in users of methylprednisolone compared to prednisolone. The exposure is prescriptions of methylprednisolone or prednisolone tablets and the primary outcome is heart failure hospitalizations within the following 6 months, i.e. acute contacts with secondary or tertiary health care resulting in a primary diagnosis of heart failure. Secondary outcomes include broader heart failure diagnoses and the initiation of loop diuretics. Data preparation includes an initial observation period of 2 years, inclusion criteria such as age, corticosteroid formulation types / dosages and prescription codes, as well as removal of duplicate prescriptions and measures to reduce potential carry-over effects.

ELIGIBILITY:
1. Individuals aged < 18 years in January 2008 will be excluded
2. Analyses will be restricted to tablets, as prednisolone is only available in this form.
3. To allow for equipotent dose comparisons, we will focus only on 4 mg and 16 mg methylprednisolone and their counterparts in prednisolone at 5 mg and 20 mg, respectively. Patients with other doses will be excluded.
4. To facilitate comparisons of treatments prescribed for similar conditions, we will only include prescriptions with an International Classification of Diseases, 10th Edition (ICD10) or International Classification of Primary Care, 2nd Edition (ICPC2) refund code.
5. Patients with prescriptions for diagnosis codes including palliative care, cancer symptoms, medical complications, and organ transplants will be excluded. This exclusion aims to reduce the inherent heterogeneity within these groups, allowing for a more comparable baseline risk.
6. An initial 2-year observational period, spanning from January 2008 to December 2009, will be used to establish comorbidities. Accordingly, only prescriptions of methylprednisolone or prednisolone dispensed from January 2010, onward, will be eligible for analyses.
7. To minimize the risk of carry-over effects, we will exclude all prescriptions prescribed < 6 months after another prescription for a corticosteroid. Accordingly, the same patient can contribute data on several treatment courses, provided that there was > 6 months since the last prescription was dispensed (See section 7 for justification for why a 6-month interval was chosen).
8. Duplicate prescriptions (same date, drug and dosage) will be kept in the analyses as a single treatment course. Cases of duplicate prescriptions on the same date, but where the drug or dosage is different will be excluded.
9. Baseline of the treatment course will be defined as the date when the prescription of either methylprednisolone or prednisolone was dispensed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This registry-based study will include data from the nationwide Norwegian Cardio-Rheuma Registry (NCRR) that encompasses the entire Norwegian adult population over a ten-year period from January 2008 to December 2017.
Sampling Method: Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Acute heart failure | 6 months
  Acute hospital contact (secondary or tertiary healthcare facilities) where the patient was given a primary diagnosis code for heart failure (ICD10 code i50*) at discharge (dead or alive).

SECONDARY OUTCOMES:
Any heart failure diagnosis, acute or elective | 6 months
  Any contact (acute or elective) with secondary or tertiary healthcare facilities where a primary diagnosis of heart failure is recorded
Newly prescribed loop diuretics or any increase in doses | 6 months
  Initiation of newly prescribed loop diuretics or any increase in doses of loop diuretics
A combination of outcome 2 and 3 | 6 months
  ny contact (acute or elective) with secondary or tertiary healthcare facilities where a primary diagnosis of heart failure is recorded, and / or initiation of newly prescribed loop diuretics or any increase in doses of loop diuretics.

OTHER OUTCOMES:
Only individuals with existing heart failure | 6 months
  Analyses of all primary and secondary outcomes including only individuals with existing heart failure
Only individuals with existing heart failure or atherosclerotic cardiovascular disease | 6 months
  Analyses of all primary and secondary outcomes including only individuals with existing heart failure or established atherosclerotic cardiovascular disease
Only individuals with at least 3 comorbidities | 6 months
  Analyses of all primary and secondary outcomes including only individuals with at least three of the following:
  * Atherosclerotic cardiovascular disease (coronary, cerebral and peripheral artery disease)
  * Chronic kidney disease
  * Diabetes (type 1 and 2)
  * Hypertension
  * Heart failure
  * Chronic obstructive pulmonary disease
  * Use of lipid-lowering drugs

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-10-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT06468007/SAP_001.pdf